CLINICAL TRIAL: NCT05203276
Title: A Prospective, Multi-center, Single-arm Exploratory Clinical Study of Envafolimab Combined With Endostar in the First-line Treatment of Driver Gene-negative Advanced Non-small Cell Lung Cancer With PD-L1 Positive Expression
Brief Title: Envafolimab Combined With Endostar in the First-line Treatment of Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endouble
Record Dates: First submitted 2022-01-06; First posted 2022-01-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Lung Neoplasms
Keywords: Envafolimab; Endostar; NSCLC; PD-L1
MeSH Terms: conditions — Lung Neoplasms | interventions — envafolimab; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab+ Endostar Group (Experimental): Envafolimab（300mg，SC，Q3W，d1） Endostar（210mg，CIV 72h，Q3W，d1-3）
  Interventions: Drug: Envafolimab; Drug: Endostar

INTERVENTIONS:
Drug: Envafolimab — 300mg，SC，Q3W，d1
  Other Names: EN WEI DA
Drug: Endostar — 210mg，CIV，Q3W，d1-3
  Other Names: ENDO

SUMMARY:
To evaluate the efficacy and safety of envafolimab combined with endostar in the first-line treatment of advanced Non-small Cell Lung Cancer With PD-L1 positive expression

DETAILED DESCRIPTION:
Endostar indication: ENDOSTAR + NP chemotherapy regimen is used to treat Stage III/IV NSCLC patients either untreated or pretreated. This indication is based on a completed multi-center Phase III clinical trial.

Envafolimab indication: Envolimab is the world's first subcutaneous injection of PD-L1 monoclonal antibody.Suitable for adult patients with advanced solid tumors with unresectable or metastatic microsatellite highly unstable (MSI-H) or mismatch repair gene defects (dMMR).

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily joins the study, can complete the signing of the informed consent form, and has good compliance;
2. Age from 18 to 80 years old (when signing the informed consent form), both male and female;
3. According to the 8th edition of the TNM staging classification of lung cancer by the International Association for the Research of Lung Cancer and the American Joint Committee on Cancer Classification, the driver gene (EGFR/ALK/ROS1) is negative and untreated patients with stage IIIB to IV NSCLC;
4. Archived tumor tissue samples or newly obtained (without anti-tumor treatment since the biopsy) core or tumor lesions (not receiving radiotherapy) excised biopsy tissue have been provided. Formalin-fixed and paraffin-embedded (FFPE) tissue blocks are better than sections. The newly obtained biopsy tissue is better than the archived tissue, and the tissue samples are tested by immunohistochemistry for PD-L1 ≥ 1%;
5. According to the evaluation criteria for the efficacy of solid tumors (RECIST Version 1.1), there is at least one imaging measurable lesion; that is, in CT or MRI detection, the longest diameter of a single lesion is ≥10mm, or the lymph node is pathologically enlarged, and a single lymph node is scanned by CT Short diameter ≥15mm;
6. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0-1;
7. The expected survival period is ≥3 months;
8. Newly treated patients who have not received systematic anti-tumor therapy, including radiotherapy and chemotherapy, targeted and immunotherapy, or patients who relapse after follow-up after adjuvant chemotherapy for more than 6 months;
9. With sufficient organ and bone marrow function, the laboratory test values within 7 days before entry into the group meet the following requirements (no blood components, cell growth factors, albumin and other corrective treatment drugs are allowed within the first 14 days of obtaining laboratory tests ),details as follows:

1) Blood routine: absolute neutrophil count (ANC) ≥1.5×109/L, platelet (PLT) ≥75×109/L, hemoglobin (HGB) ≥90 g/L (no blood transfusion or no red blood cells within 14 days) Genin-dependent); 2) Liver function: serum total bilirubin (TBIL) ≤2 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤5 times ULN, serum Albumin ≥28 g/L; Alkaline phosphatase (ALP) ≤5×ULN; 3) Renal function: Serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥50 mL/min (using the standard Cockcroft-Gault formula): urine routine results show urine protein <2+; urine routine testing at baseline Patients who show urine protein ≥2+ should be collected for 24 hours and the quantification of 24-hour urine protein should be less than 1g; 4) Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, as long as the INR is within the intended use range of anticoagulant drugs; 10. For female subjects of childbearing age, a urine or serum pregnancy test should be performed 3 days before receiving the first study drug administration and the result is negative; 11. It is necessary to provide tissue samples for biomarker (such as PD-L1) analysis, preferably newly obtained tissues. Patients who cannot provide newly obtained tissues can provide 3-5μm-thick paraffin sections of tissues that are archived and saved within 2 years before enrollment. 5-8 sheets.

Exclusion Criteria:

1. Imaging (CT or MRI) shows that the tumor has invaded large blood vessels or those who are judged to be very likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study;
2. Currently participating in interventional clinical research treatment, or receiving treatment with other research drugs or research devices within 4 weeks before the first administration;
3. Received Chinese patent medicines with anti-tumor indications or immunomodulatory drugs (thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration, or received major surgery within 3 weeks before the first administration;
4. There are active hemoptysis, active diverticulitis, abdominal abscess, gastrointestinal obstruction and peritoneal metastasis that require clinical intervention;
5. Regardless of the severity, patients with any signs of bleeding or medical history; patients with any bleeding or bleeding event ≥ CTCAE level 3 within 4 weeks before enrollment, unhealed wounds, ulcers or fractures;
6. Grade III-IV congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmia;
7. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, occurred within 6 months before being selected for treatment;
8. Known to have allergic reactions to the drug in this study;
9. Patients who require long-term systemic use of corticosteroids. Patients who require intermittent use of bronchodilators, inhaled corticosteroids, or local injections of corticosteroids due to COPD and asthma can be included in the group;
10. Symptomatic central nervous system metastasis. Patients with asymptomatic brain metastases or brain metastases with stable symptoms after treatment can participate in this study as long as they meet all the following criteria: there are measurable lesions outside the central nervous system; no midbrain, pons, cerebellum, meninges, Medulla oblongata or spinal cord metastasis; maintain a clinically stable state for at least 2 weeks; stop hormone therapy 3 days before the first dose of study drug;
11. There is an active infection that needs to be treated or systemic anti-infective drugs have been used within one week before the first administration;
12. Before starting treatment, have not fully recovered from toxicity and/or complications caused by any intervention (ie, ≤ Grade 1 or reached baseline, excluding fatigue or hair loss);
13. Known human immunodeficiency virus (HIV) infection history (ie HIV 1/2 antibody positive);
14. Untreated active hepatitis B (defined as HBsAg positive and the number of copies of HBV-DNA detected at the same time is greater than the upper limit of the normal value of the laboratory department of the research center);

Note: Hepatitis B subjects who meet the following criteria can also be included in the group:

1. The HBV viral load before the first administration is less than 1000 copies/ml (200 IU/ml), and the subject should receive anti-HBV treatment during the entire study chemotherapy drug treatment period to avoid viral reactivation;
2. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-), there is no need to receive preventive anti-HBV treatment, but close monitoring of virus reactivation is required.

15. Active HCV infected subjects (HCV antibody-positive and HCV-RNA level is higher than the lower limit of detection); 16. Live vaccine has been vaccinated within 30 days before the first administration (cycle 1, day 1); Note: It is allowed to receive inactivated virus vaccine for seasonal influenza within 30 days before the first administration; however, it is not allowed to receive live attenuated influenza vaccine for intranasal administration.

17. Pregnant or lactating women; 18. The medical history or disease evidence, abnormal treatment or laboratory test values that may interfere with the test results, prevent the subjects from participating in the study, or the investigator believes that it is not suitable for inclusion in the group. The investigator believes that there are other potential risks and is not suitable for participation this research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  The proportion of patients whose tumor volume has reduced to a predetermined value and can maintain the minimum time limit
Number of participants with adverse events as a measure of safety and tolerability | up to 24 months
  From randomization until death (up to 24 months)

SECONDARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Progression-free survival
DCR | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate
OS | From randomization until death (up to 24 months)
  Overall survival
DOR | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Jiang, Doc, Study Chair — The First People's Hospital of Lianyungang
Locations (1):
- The First People'S Hospital of Lainyungang, Lianyungang, Jiangsu, China

REFERENCES:
- [Background] Fukumura D, Kloepper J, Amoozgar Z, Duda DG, Jain RK. Enhancing cancer immunotherapy using antiangiogenics: opportunities and challenges. Nat Rev Clin Oncol. 2018 May;15(5):325-340. doi: 10.1038/nrclinonc.2018.29. Epub 2018 Mar 6. PMID 29508855
- [Background] Hockenhull K, Ortega-Franco A, Califano R. Pembrolizumab plus platinum-based chemotherapy for squamous non-small cell lung cancer: the new kid on the block. Transl Lung Cancer Res. 2021 Sep;10(9):3850-3854. doi: 10.21037/tlcr-20-715. No abstract available. PMID 34733633
- [Background] Borghaei H, Langer CJ, Paz-Ares L, Rodriguez-Abreu D, Halmos B, Garassino MC, Houghton B, Kurata T, Cheng Y, Lin J, Pietanza MC, Piperdi B, Gadgeel SM. Pembrolizumab plus chemotherapy versus chemotherapy alone in patients with advanced non-small cell lung cancer without tumor PD-L1 expression: A pooled analysis of 3 randomized controlled trials. Cancer. 2020 Nov 15;126(22):4867-4877. doi: 10.1002/cncr.33142. Epub 2020 Sep 11. PMID 32914866
- [Result] Jiang XD, Dai P, Wu J, Song DA, Yu JM. Effect of recombinant human endostatin on radiosensitivity in patients with non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):1272-7. doi: 10.1016/j.ijrobp.2011.09.050. Epub 2011 Nov 16. PMID 22099051